CLINICAL TRIAL: NCT00185809
Title: Scintigraphic Assessment of I- Transport in Metastatic Breast Cancer and Evaluation of I31I Ablative Therapy: (Part I) Radioiodide Imaging Study
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Irene L. Wapnir, Stanford University School of Medicine
Other Study IDs: BRSMTS0002; 75632; BRSMTS0002; NCT00185809; NIH
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Archival tissue blocks and blood

SUMMARY:
The purpose of this study is to examine breast cancers that express the protein (NIS) that may be found in malignant breast tissues and to evaluate proteins found in blood and their relationship to NIS, to test whether iodide can be concentrated by breast cells to possibly treat some breast cancers with radioactive iodine, and to calculate the amount of radioactive iodine entering breast cancer cells, how long your cancer retains the agent as well as how much is taken up by other organs, particularly the thyroid gland.

DETAILED DESCRIPTION:
To demonstrate iodide uptake capacity of breast cancer metastases by imaging women with iodide radioisotope (123I) and calculating potential ablative dose of radioactive iodide (131I).

ELIGIBILITY:
Inclusion Criteria:- Only women diagnosed with breast cancer

* 18 years of age or older
* From whom informed consent can be obtained
* Patient is able to provide a fluid (e.g. cyst fluid)
* Patient with blood test that shows protein may allow iodide to accumulate in breast tissue
* Patient who's breast cancer cells accumulated I123 and held on to it for 24 hours Exclusion Criteria:- Males
* Children

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligibility criteria include histological proof of invasive breast cancer and current radiological evidence of metastatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2000-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene L. Wapnir, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States